CLINICAL TRIAL: NCT00834470
Title: Is Atropine Needed With Ketamine Sedation?
Brief Title: Adjunctive Atropine During Ketamine Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Hee Lee, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Atropine-01
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Conscious Sedation
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atropine (Experimental): Atropine 0.01mg/kg IV
  Interventions: Drug: Atropine
- Normal saline (Placebo Comparator): Same volume of atropine
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — Ketamine 2mg/kg IV + Atropine 0.01mg/kg or Same volume of Normal saline

SUMMARY:
* Ketamine seems an obvious choice in the setting of an emergency department
* Ketamine leads to increased production of salivary and tracheal secretions
* Antisialagogues(atropine)therefore have been recommended as a routine adjunct
* We compare atropine with placebo as an adjunct to ketamine sedation in children undergoing primary closure of lacerated wound

DETAILED DESCRIPTION:
The degree of secretion was significantly less in the atropine group compared with the control group at the end of the procedure (VAS score: 16.5 ± 9.9 vs. 27.0 ± 15.9, atropine vs. control, p = 0.00). The change in the degree of secretion between the start and end of the procedure was significantly greater in the atropine group than in the control group (p = 0.00) (Fig. 2). However, the frequency of hypersalivation as predefined (VAS score ≥50) did not differ between the groups (p = 0.06).

The only complication that differed significantly between the two groups was tachycardia (p > 0.05). Complications such as aspiration, laryngospasm, and apnea were not documented in the hospital. There were fewer interventions for hypersalivation in the atropine group, but the difference was not significant (p > 0.05). As interventions, O2 administration and endotracheal intubation were not needed. After discharge, the control patients tended to have more complaints of nausea, vomiting, and ataxia, although the difference was not significant (p > 0.05) Heart rate was increased significantly in the atropine group (p = 0.00). The frequency of tachycardia according to patient age was also significantly higher in the atropine group than in the control group (p = 0.00)

ELIGIBILITY:
Inclusion Criteria:

* Pediatric lacerated patients

Exclusion Criteria:

* Contraindication of ketamine or atropine

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hypersalivation(VAS) | During procedure

SECONDARY OUTCOMES:
Sedation scale | before, during procedure, before discharge
Pain scale | before, during procedure, before discharge
Complication | during procedure and bedore discharge and 1day after discharge
Satisfaction of parents and clinicians | before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hee Lee, Professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kye YC, Rhee JE, Kim K, Kim T, Jo YH, Jeong JH, Lee JH. Clinical effects of adjunctive atropine during ketamine sedation in pediatric emergency patients. Am J Emerg Med. 2012 Nov;30(9):1981-5. doi: 10.1016/j.ajem.2012.04.030. Epub 2012 Jun 28. PMID 22748697